CLINICAL TRIAL: NCT00673621
Title: A Phase 1, Open-Label, Controlled Clinical Trial to Evaluate Pharmacokinetics After Administration of Technosphere® Insulin Inhalation Powder Alone and With Salbutamol (Albuterol) and/or After Methacholine Challenge Testing in Subjects With Asthma Versus Matched Healthy Subjects Without Asthma
Brief Title: A Study Designed to Determine if the Pharmacokinetic Disposition of Inhaled Insulin Exposure is the Same for Asthmatics and Non-asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-113
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Asthma; Diabetes Mellitus
Keywords: Asthmatics and non-asthmatic male and female subjects
MeSH Terms: conditions — Asthma; Diabetes Mellitus | interventions — Albuterol; Methacholine Chloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Technosphere Insulin Inhalation Powder; Drug: Salbutamol (Albuterol); Drug: Methacholine chloride

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder — 3.0 of human insulin. single dose cartridges filled with 5 or 10 mg of Technosphere Inhalation Powder, containing 15 or 30 u of insulin
Drug: Salbutamol (Albuterol) — 2 puff = 200 mcg total dose
Drug: Methacholine chloride — 5mls of methacholine; diluent sodium chloride 0.9%; formulation methacholine chloride in sodium chloride 0.9%

SUMMARY:
This study will compare the rate and extent of absorption of TI Inhalation Powder in subjects with asthma and subjects with normal lung function. 24 eligible subjects will be enrolled into the treatment phase of the trial.

DETAILED DESCRIPTION:
Visit 1 screening will determine eligibility and obtain informed consent. At visit 2, 3 and 4 subjects inhale 1 dose of 45U TI Inhalation Powder. At visit 3 subjects inhale 2 puffs (200mcg) Albuterol prior to dosing. Only asthmatic subjects undergo visit 4 where a methacholine challenge test (MCT) is performed followed by inhalation of Albuterol then administration of TI Inhalation Powder. Each visit's dosing will occur during a hyperinsulinemic euglycemic clamp. Visit 5 is the follow up visit.

ELIGIBILITY:
Inclusion Criteria:

Non smoking male and female subjects = 18 and = 55 years of age with BMI = 34 kg/m2 Fasting blood glucose (FBG) < 110 mg/dL (6.1 mmol/L). Written informed consent Asthmatic Subjects: Clinical diagnosis of asthma along with defined reversibility from pre- to post-bronchodilator spirometry.

Pulmonary Function Testing for Asthmatic subjects: FEV1 > 70% (NHANES III), TLC >70% (ITS), Dlco >80% (Miller) Non-asthmatic healthy subjects: FEV1 > 80% (NHANES III), FEV1/FVC > LLN (NHANES), TLC >80% (ITS), Dlco >80% (Miller), no significant improvement from pre- to post-bronchodilator spirometry.

Exclusion Criteria:

Unable and/or unlikely to comprehend how to use the investigational device in this study or to follow study instructions Change in asthma therapeutic regimen from Screening through visit 5 Exacerbation of asthma within 8 weeks prior to Screening History of diabetes mellitus Previous exposure to any inhaled insulin product other than TI inhalation Powder or similar formulation Inability to perform PFT maneuvers meeting recommended American Thoracic Society (ATS) standards of acceptability and repeatability criteria Any clinically important pulmonary disease Major organ system diseases including seizures, heart failure, uncontrolled hypertension, cancer within the past 5 years, aneurysm, liver disease, anemia or autoimmune disorder Clinically significant abnormalities on screening laboratory evaluation Female subjects who are pregnant, lactating, or planning to become pregnant during the clinical trial period or not practicing adequate birth control

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
AUCF 0-360 min of serum insulin | 0-360 min

CONTACTS AND LOCATIONS:
Overall Officials: Anders H. Boss, Study Chair — Mannkind Corporation
Locations (2):
- United Kingdom (2):
  - Medicines Evaluation Unit (MEU), Manchester, England
  - ICON Development Solutions, Manchester